CLINICAL TRIAL: NCT04252287
Title: Canagliflozin: Impact on Health Status, Quality of Life, and Functional Status in Heart Failure
Brief Title: A Study on Impact of Canagliflozin on Health Status, Quality of Life, and Functional Status in Heart Failure
Acronym: CHIEF-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108750; 28431754HFA3002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canagliflozin 100 mg (Experimental): Participants will be administered 100 milligram (mg) immediate-release, over-encapsulated tablets (as a capsule) orally once daily for 12 weeks.
  Interventions: Drug: Canagliflozin 100 mg
- Placebo (Placebo Comparator): Participants will be administered matching placebo capsules orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 100 mg — Participants will receive 100 mg immediate-release, over-encapsulated tablets (as a capsule) orally once daily.
  Other Names: JNJ-28431754; INVOKANA
  Arms: Canagliflozin 100 mg
Drug: Placebo — Participants will receive matching placebo capsules orally once daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the superiority of the effectiveness of canagliflozin 100 milligram (mg) daily versus placebo in participants with symptomatic heart failure (HF) in improving the overall Kansas City Cardiomyopathy Questionnaire (KCCQ) Total Symptom Score (TSS).

ELIGIBILITY:
Inclusion Criteria:

- Have clinically stable symptomatic heart failure (HF) (heart failure with reduced ejection fraction [HFrEF] and heart failure with preserved ejection fraction [HFpEF]): (A) For HFrEF: (a) ejection fraction (EF) less than or equal to (<=) 40 percent (%) and (b) a primary diagnosis of HF OR 2 medical visits (including virtual) with a HF diagnosis code in any position in the past 18 months (B) For HFpEF: (a) EF greater than (>) 40%; (b) a primary diagnosis of HF OR 2 medical visits (including virtual) with a HF diagnosis code in any position in the past 18 months, AND; (C) on a loop diuretic or spironolactone or eplerenone (mineralocorticoid receptor antagonists), in the past 18 months

* Have a baseline Kansas City Cardiomyopathy Questionnaire (KCCQ) score of less than or equal to (<=) 80 prior to randomization
* Be able to read and understand English
* Possess and have sole use (example: not shared with other users) of smartphone compatible with the Fitbit device
* Willing/able to wear the Fitbit device on a regular basis for the 9-month study period

Exclusion Criteria:

* Currently taking a sodium-glucose co-transporter 2 inhibitor (SGLT2i) or within the last 3 months
* History of diabetic ketoacidosis or have type 1 diabetes mellitus (T1DM)
* Have acute decompensated HF (exacerbation of symptomatic HF) requiring intravenous diuretics, inotropes, or vasodilators within the last 4 weeks
* Have stage 4 or 5 Chronic Kidney Disease (that is, estimated glomerular filtration rate [eGFR] <30 milliliter per minute [ml/min] on dialysis) from the most recent assessment
* Have a diagnosis of hypotension within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (18):
- United States (18):
  - Mercy Clinic Cardiology - Fort Smith, Fort Smith, Arkansas
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Emory University, Atlanta, Georgia
  - St Lukes Regional Medical, Boise, Idaho
  - OSF HealthCare Cardiovascular Institute, Peoria, Illinois
  - Central Dupage Hospital, Winfield, Illinois
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - MedStar Health Research Institute, Hyattsville, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Luke's Hospital Kansas City, Kansas City, Missouri
  - Mercy Health Research, Washington, Missouri
  - Robert Wood Johnson Medical School Dept. of Medicine, Piscataway, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Thomas Spann Clinic, Corpus Christi, Texas
  - Texas Heart Institute, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Mohebi R, Jones PG, Spertus JA, Lingvay I, Lanfear DE, Gosch KL, Birmingham M, Kosiborod MN, Butler J, Januzzi JL Jr. Early Longitudinal Change in Heart Failure Health Status Following Initiation of Canagliflozin. JACC Heart Fail. 2024 Apr;12(4):711-718. doi: 10.1016/j.jchf.2024.01.005. Epub 2024 Feb 21. PMID 38385941
- [Derived] Golbus JR, Gosch K, Birmingham MC, Butler J, Lingvay I, Lanfear DE, Abbate A, Kosiborod ML, Damaraju CV, Januzzi JL Jr, Spertus J, Nallamothu BK. Association Between Wearable Device Measured Activity and Patient-Reported Outcomes for Heart Failure. JACC Heart Fail. 2023 Nov;11(11):1521-1530. doi: 10.1016/j.jchf.2023.05.033. Epub 2023 Jul 26. PMID 37498273
- [Derived] Nassif M, Birmingham MC, Lanfear DE, Golbus JR, Gupta B, Fawcett C, Harrison MC, Spertus JA. Recruitment Strategies of a Decentralized Randomized Placebo Controlled Clinical Trial: The Canagliflozin Impact on Health Status, Quality of Life and Functional Status in Heart Failure (CHIEF-HF) Trial. J Card Fail. 2023 Jun;29(6):863-869. doi: 10.1016/j.cardfail.2023.04.001. Epub 2023 Apr 10. PMID 37040839
- [Derived] Spertus JA, Birmingham MC, Nassif M, Damaraju CV, Abbate A, Butler J, Lanfear DE, Lingvay I, Kosiborod MN, Januzzi JL. The SGLT2 inhibitor canagliflozin in heart failure: the CHIEF-HF remote, patient-centered randomized trial. Nat Med. 2022 Apr;28(4):809-813. doi: 10.1038/s41591-022-01703-8. Epub 2022 Feb 28. PMID 35228753
- [Derived] Spertus JA, Birmingham MC, Butler J, Lingvay I, Lanfear DE, Abbate A, Kosiborod ML, Fawcett C, Burton P, Damaraju CV, Januzzi JL, Whang J. Novel Trial Design: CHIEF-HF. Circ Heart Fail. 2021 Mar;14(3):e007767. doi: 10.1161/CIRCHEARTFAILURE.120.007767. Epub 2021 Mar 16. PMID 33724883

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1,333 participants were screened. Of which, 476 participants were randomized in the study.
Groups:
- Placebo: Participants received placebo (matched to canagliflozin) capsule orally once daily for 12 weeks.
- Canagliflozin 100 mg: Participants received canagliflozin 100 milligrams (mg) immediate-release, over-encapsulated tablet (as capsule) orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg
Started | 238 | 238
Treated (Safety Analysis Set) (Safety analysis set included all randomized participants who received at least 1 dose of study intervention.) | 231 | 224
Completed | 207 | 209
Not Completed | 31 | 29
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Total
Number analyzed (Participants) | 231 | 224 | 455
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (13.5) | 62.9 (13.15) | 63.4 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 105 | 204
  Male | 132 | 119 | 251
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 199 | 184 | 383
  Black or African American | 30 | 35 | 65
  Asian | 1 | 1 | 2
  Other | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Kansas City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) at Week 12
Description: Change from baseline in KCCQ-TSS was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-TSS was average of domains- symptom frequency and symptom burden, and transformed to a single score which ranged from 0 (worst) to 100 (the best possible status), where the higher score reflected better health status.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized participants who had received at least one dose of study intervention/medication and had at least one post-baseline KCCQ measurement. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 206 | 208
Score on a scale | 4.9 (1.27) | 9.2 (1.27)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority; p = 0.016, ANCOVA; LS mean difference = 4.3, 95% CI 2-sided [0.8 to 7.8]

2. Secondary Outcome: Change From Baseline in Total Daily Step Count at Week 12
Description: Change from baseline in total daily step count at Week 12 was reported in this outcome measure. The number of steps taken per day was measured using a step activity monitor at baseline and throughout the study. Step count was measured from the Fitbit device data. The Fitbit app on the participant's phone collected all data from the Fitbit device. A negative change from baseline indicated a decrease in the number of daily steps.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who had received at least one dose of study intervention/medication and had at least one post-baseline KCCQ measurement. Here, N (Overall number of participants analyzed) signifies participants evaluated for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Daily step count
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 208 | 205
Daily step count | -74.9 (112.85) | -45.1 (113.78)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Test type: Superiority; p = 0.852, ANCOVA; LS mean difference = 29.8, 95% CI 2-sided [-284.4 to 344.1]

3. Secondary Outcome: Change From Baseline in KCCQ Individual Domain Scores (Physical Limitation and Quality of Life) at Week 12
Description: Change from baseline in KCCQ physical limitation score and KCCQ quality of life score were reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 (worst) and 100 (the best possible status), where the higher score reflected better health status.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who had received at least one dose of study intervention/medication and had at least one post-baseline KCCQ measurement. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants with available data for each specified category.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 206 | 208
Score on a scale
  KCCQ-Physical Limitation: number analyzed (Participants) | 206 | 204
  KCCQ-Physical Limitation | 4.8 (1.26) | 7.8 (1.27)
  KCCQ-Quality of Life | 9.1 (1.40) | 12.4 (1.41)

4. Secondary Outcome: Change From Baseline in KCCQ Clinical Summary Score at Week 12
Description: Change from baseline in KCCQ-clinical summary score was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ-clinical summary score was average of domains- physical limitation and total symptoms (average of symptom frequency and symptom burden), and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Time Frame: Baseline, Week 12
Population: FAS included all randomized participants who had received at least one dose of study intervention/medication and had at least one post-baseline KCCQ measurement. Here, N (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 206 | 208
Score on a scale | 4.7 (1.16) | 8.5 (1.17)

5. Secondary Outcome: Change From Baseline in KCCQ Overall Summary Score at Week 12
Description: Change from baseline in KCCQ-overall summary score was reported. KCCQ was a 23-item, self-administered questionnaire that measure the participant's perception of their health status, including their heart failure (HF) symptoms, impact on physical and social function and how their HF impacts the quality of life. KCCQ quantifies 7 domains: physical limitations (6 items), symptom stability (1 item), symptom frequency (4 items), symptom burden (3 items), self-efficacy (2 items), quality of life (3 items) and social limitations (4 items). Scores were generated for each domain and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status. KCCQ- overall summary score was average of domains- physical limitation, total symptoms (average of symptom frequency and symptom burden), quality of life, and social limitation, and transformed to a single score which ranged from 0 (worst) -100 (the best possible status), where the higher score reflected better health status.
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 206 | 208
Score on a scale | 6.2 (1.18) | 9.5 (1.18)

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 9 months; serious adverse events and other adverse events: Up to 30 days after end of treatment (up to 4 months)
Description: Safety analysis set included all randomized participants who received at least 1 dose of study intervention.
Arm/Group | Placebo | Canagliflozin 100 mg
All-Cause Mortality (participants affected / at risk) | 5/231 | 3/224
Serious Adverse Events (participants affected / at risk) | 36/231 | 33/224
Other Adverse Events (participants affected / at risk) | 0/231 | 0/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=231) | Canagliflozin 100 mg (N=224)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 4
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 2
Sudden cardiac death (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 4
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 2 | 0
Weight increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Bell's palsy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac operation (Surgical and medical procedures) | 0 | 1
Implantable defibrillator replacement (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04252287/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT04252287/SAP_003.pdf